CLINICAL TRIAL: NCT00606125
Title: Phase I Study With Sorafenib in Combination With Carboplatin and Paclitaxel to Evaluate the Safety and Pharmacokinetics of This Combination in Patients With Solid Tumors
Brief Title: Sorafenib/ Carboplatin/ Paclitaxel in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11988
Record Dates: First submitted 2008-01-21; First posted 2008-02-01 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms
Keywords: Chemotherapy; Solid Tumors; Sorafenib; Carboplatin; Paclitaxel
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — The purpose of this study is to: 1)evaluate how your body reacts to sorafenib when taken daily in combination with paclitaxel and carboplatin, 2) measure your blood levels of sorafenib, paclitaxel and carboplatin at specific times after taking the medication, and 3) to determine the safety of sorafenib.

SUMMARY:
The purpose of this study is to:

1. Evaluate how the body reacts to sorafenib when taken daily in combination with paclitaxel and carboplatin,
2. Measure the blood levels of sorafenib, paclitaxel and carboplatin at specific times after taking the medication, and
3. To determine the safety of sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years
* Histological or cytological documentation of cancer, except non small cell lung cancer
* ECOG Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* No more than two prior chemotherapy regimens
* Adequate bone marrow, liver and renal function as assessed by the following:

  * Hemoglobin > or equal to 9.0 g/dL
  * Absolute neutrophil count (ANC) > or equal to 1,500/mm3
  * Platelet count > or equal to 100,000/mm3
  * Total bilirubin < or equal to 1.25 times the ULN
  * ALT and AST < or equal to 2.5 x ULN
  * PT-INR/PTT < 1.5 x ULN (Patients who are being prophylactically anti coagulated with an agent such as coumadin or low molecular weight heparin or therapeutically anticoagulated with LMWH will be allowed to participate provided that they meet these criteria; in addition, these patients must be monitored at appropriate intervals throughout study)
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation, including the 30 day period after last study drug dosing. The investigator should advise the patient regarding adequate means of contraception.
* Serum creatinine < or equal to 1.5 x upper limit of normal
* Ability to understand and willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* Clinically evident congestive heart failure > NYHA Class 2 (See Appendix 10.4)
* Serious cardiac arrhythmias (for example requiring anti-arrhythmics)
* Myocardial infarction or symptomatic coronary artery disease (severe or unstable angina) within 6 months prior to screening
* Active clinically serious infections (> Grade 2 NCI-CTC)
* Patients with history of brain metastases are eligible as long as the metastasis has been treated with either stereotactic or whole brain radiation, stereotactic gamma-knife radiosurgery or neurosurgery, patient does not require ongoing treatment with dexamethasone, the patient is not on anticoagulant therapy and whose radiographic imaging is stable ≥ 4 weeks from start of treatment. Time from brain metastasis treatment to first study treatment must meet the following criteria:

  * Stereotactic or whole brain radiation, stereotactic gamma-knife radiosurgery ≥ 4 weeks from first study treatment
  * Neurosurgery ≥ 24 weeks from first study treatment
  * Brain biopsy ≥ 12 weeks from first study treatment
* History of organ allograft
* Uncontrolled seizure disorder. Use of cytochrome P450 enzyme-inducing antiepileptic drugs (phenytoin, carbamazepine or phenobarbital) is not allowed
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management
* Known human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Peripheral neuropathy > or equal to Grade 2
* Thrombotic or embolic events (such as transient ischemic attacks, myocardial infarction, pulmonary embolus), within 6 months prior to Screening
* Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first study treatment
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first study treatment
* Evidence or history of bleeding diathesis or coagulopathy
* Serious, non-healing wound, ulcer, or bone fracture
* Patients undergoing renal dialysis
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study treatment
* Previous cancer EXCEPT cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors [Ta and Tis] or any cancer curatively treated > 3 years prior to first study treatment
* Non small cell lung cancer
* Ongoing substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Pregnant or breast-feeding patients.
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study
* Any condition that impairs patient's ability to swallow whole pills
* Any malabsorption condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety and pharmacokinetics of the three agents: sorafenib administered daily, without a break in dosing, in combination with carboplatin and paclitaxel, administered every 3 weeks | 2 years

SECONDARY OUTCOMES:
To determine the safety profile and pharmacokinetics of oral sorafenib daily in combination with every 3-weekly carboplatin and paclitaxel. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - New Haven, Connecticut
  - San Antonio, Texas